CLINICAL TRIAL: NCT04190836
Title: Adherence to Self-managed Exercises for Patients With Persistent Subacromial Pain: A Feasibility Study for the Ad-Shoulder Trial
Brief Title: Self-Management for Persistent Subacromial Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Oslo University Hospital (Other); Keele University (Other); National Institute of Occupational Health (Unknown); Diakonhjemmet Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/355
Record Dates: First submitted 2019-11-18; First posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Shoulder Pain Chronic
Keywords: Shoulder pain; Persistent pain; Self-management; Exercise
MeSH Terms: conditions — Shoulder Pain; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-Managed Exercise Strategy (Experimental)
  Interventions: Behavioral: Self-Managed Exercise Strategy

INTERVENTIONS:
Behavioral: Self-Managed Exercise Strategy — The intervention is a personalised supported self-management intervention which emphasises dynamic, progressively loaded exercises for the shoulder. The intervention consisted of 1-5 individual sessions provided over 3 months, with a duration of 1 hour for the first session and 45 minutes for the following. The participants will have the opportunity to contact the physiotherapist by phone, text message or e-mail for advice during the treatment period (12 weeks). The personalised supported self-management intervention will be based on the components of the self-management framework, provided by Lorig and Holman (2003). The five self-management skills and the operationalization of these will be described when publishing the study. For specific content reporting of the self managed exercises we will follow the Consensus on Exercise Reporting Template.

SUMMARY:
Physiotherapy-led exercises is the first line treatment for patients with subacromial pain. However, current evidence report that most treatment programmes only show a short-term benefit. There seem to be a potential for enhancing the effectiveness of exercise interventions by improving adherence to self-managed exercises, but there is lack of knowledge about adherence to exercise programmes in shoulder pain. Before conducting a planned randomised controlled trial on the clinical effectiveness of an intervention focusing on adherence to a self-managed exercise strategy (the Ad-Shoulder intervention), it is necessary to run a feasibility study in order to establish whether such a resource-demanding trial is worthwhile. Feasibility studies are designed to answer the key question "Can it work?" The main objectives of the present study was to assess the feasibility in terms of recruitment capability, data collection procedures and acceptability of the Ad-Shoulder intervention in patients with subacromial pain receiving treatment in primary or secondary health care.

ELIGIBILITY:
Inclusion Criteria:

* Pain located to the upper arm
* Had previously received conservative treatment due to subacromial pain
* Still seek primary or secondary care during the past 6 months

Exclusion Criteria:

* Frozen shoulder diagnosis (<50% external rotation compared to contralateral side)
* Patients who have received surgical treatment due to shoulder problems
* Pregnant patients
* Patients with insufficient Norwegian language skills
* Serious psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 3 months
  How many people that were eligible and how many people that were recruited per week
Follow-up rate | 3 months
  Determine the follow-up rate - measured by the percentage of participants who were followed up successfully until the three months follow-up
Actigraph assessment of physical activity | 3 months
  Feasibility of Actigraph assessment of physical activity - measured by percentage of participants with valid data at Week 0, Week 6 and 3 months
Adherence | 3 months
  Determine whether the patients adhere with the self-managed exercises - measured by self-reported exercise log book
Fidelity | 3 months
  Determine whether the therapists delivered the intervention as planned - measured by assessing the therapists' log book
Adverse events | 3 months
  Determine number and nature of adverse events via self-report questionnaire

SECONDARY OUTCOMES:
Shoulder pain and disability index (SPADI) | 3 months
  SPADI is a self-reported questionnaire for patients with shoulder pain. The questionnaire consists of 13 questions divided into two domains: pain (five items) and function (eight items) and scored on a numerical scale 0 (best) to 10 (worst) with a score range from 0 to 100 points
Patient Specific Function Scale (PSFS) | 3 months
  PSFS is a patient specific outcome measure where the patient is asked to name three activities which the patient find challenging or are not able to do because of their shoulder pain. Patients rate their ability to complete the activities on a 11-point scale at a level experienced prior to injury or change in functional status. "0" represents "unable to perform" and "10" represents "able to perform at prior level".
Numeric Pain Rating Scale (NPRS) | 3 months
  Pain intensity during the last week was measured using the NPRS (ranging from 0 = no pain, 10 = the most intense pain imaginable). Repeated measures: During a one week pre-treatment phase (A), 3 times. During the 12 week treatment phase (B): collected twice every week. During a one week post-treatment phase (A): 3 times
Pain self-efficacy 2-item short form (PSEQ-2 item) | 3 months
  Measured using a 2-item questionnaire by asking the patients' how confident they are doing some form of work and to live a normal lifestyle at present, despite the pain (ranging from 0 = not at all confident, 6 = completely confident). Repeated measures: During a one week pre-treatment phase (A), 3 times. During the 12 week treatment phase (B): collected twice every week. During a one week post-treatment phase (A): 3 times
Self-efficacy | 3 months
  Measured using one modified question from the Musculoskeletal Health Questionnaire: "How confident have you felt about managing your shoulder pain by yourself (responses were not at all confident, slightly, moderately, very and extremely)? Repeated measures: During a one week pre-treatment phase (A), 3 times. During the 12 week treatment phase (B): collected twice every week. During a one week post-treatment phase (A): 3 times
Working Ability Index | 3 months
  Work ability will be measured on a 11-point scale (0 = Can not work at all, 10 = working ability is best right now)
EQ-5D-5L | 3 months
  Generic health-related quality of life will be assessed by the EQ-5D. It evaluates 5 dimensions: mobility, self-care, activities of daily living, pain, and anxiety and/or depression. For each dimension the patient describes three possible levels of problems (none, mild-to-moderate, and severe).
Global Perceived Effect scale (GPE) | 3 months
  The patient rated perception of change at the follow-ups will be assessed on a Global Perceived Effect scale (GPE) at follow-up (52). The response alternatives were: 1 = "completely recovered", 2 = "much improved", 3 = "slightly improved", 4 = "no change", 5 = "slightly worse", 6 = "much worse", and 7 = "worse than ever".
Bergen Insomnia Scale | 3 months
  Pain-interference with sleep will be assessed by the Bergen Insomnia Scale, which consists of six items. Scoring 3 or above on at least one of the first four items and scoring 3 or above on at least one of the last two items indicate the presence of insomnia.
Kinesiophobia | 3 months
  Kinesiophobia will be assessed using one question: "How much 'fear' do you have that these complaints would be increased by physical activity? (scores range from 0 = no fear, to 10 = very much fear).
Physical activity (self-reported) | 3 months
  Physical activity will be assessed by the 3 questions from the Nord-Trondelag Health Study (HUNT) regarding frequency, intensity and duration.
Physical activity (accelerometer) | 3 months
  To objectively measure physical activity an accelerometer (AX3, 3-axis Logging Accelerometer) was used. This accelerometer provides information about movement and will enable us to objectively measure the amount of general physical activity (minutes of moderate activity). The patients will be measured for three consecutive days at baseline, at 6 weeks and at 3 months to assess changes between the three time points (Week 0, Week 6 and 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Major, MSc, Study Chair — Oslo Metropolitan University; Yngve Røe, PhD, Principal Investigator — Oslo Metropolitan University; Margreth Grotle, PhD, Study Chair — Oslo Metropolitan University; Chris Littlewood, PhD, Study Chair — Keele University; Dagfinn Matre, PhD, Study Chair — National Institute of Occupational Health, Norway; Heidi V Gallet, MSc, Study Chair — Diakonhjemmet Hospital; Hege Bentzen, PhD, Study Director — Oslo Metropolitan University
Locations (2):
- Norway (2):
  - Diakonhjemmet Hospital, Oslo
  - Oslo Metropolitan University, Oslo

REFERENCES:
- [Derived] Major DH, Grotle M, Littlewood C, Brox JI, Matre D, Gallet HV, Roe Y. Adherence to self-managed exercises for patients with persistent subacromial pain: the Ad-Shoulder feasibility study. Pilot Feasibility Stud. 2021 Jan 25;7(1):31. doi: 10.1186/s40814-021-00767-6. PMID 33494821